CLINICAL TRIAL: NCT03061084
Title: Long Term Assessment and Outcome of Adult Patients With Congenital Genitourinary Abnormalities.
Brief Title: Prospective Cohort of Transitional Urology Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rose Khavari, M.D., Principal Investigator, The Methodist Hospital Research Institute
Other Study IDs: Pro00012924
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Spina Bifida; Myelomeningocele; Meningocele; Bladder Exstrophy; Genitourinary Congenital Anomalies; Cloacal Exstrophy
Keywords: Spina Bifida, Neurogenic bladder, Myelomeningocele
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele; Meningocele; Bladder Exstrophy; Urogenital Abnormalities; Cloacal Exstrophy; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A transitional Urology database was created in parallel with National Spina Bifida registry to follow patients with complex congenital urogenital anomalies and be able to prospectively evaluate them. The investigators obtained the standardized questionnaires to collect long-term data regarding patients' genitourinary status including urine and fecal continence, sexuality, fertility, and pelvic health.

DETAILED DESCRIPTION:
The care and management of pediatric patients with congenital genitourinary anomalies transitioning to adolescents and later adults is undergoing a period of profound transformation. Due to improvements in surgical and nonsurgical interventions, children with diverse congenital disease affecting the genitourinary tract are surviving into adulthood at far higher rates than in the past. As an example, up to 70-75% of children born with a myelomeningocele and consequent neurogenic bladder are living past the age of twenty. These new expectations, especially in the areas of sexual function, fertility and reproductive health, are creating previously unseen challenges for health care providers attempting to transition adolescents from pediatric to adult care. As this patient population continues to grow, the transitional process for urological care of congenital anomalies is progressively becoming a topic of vital importance.

We plan to advance adolescence clinical and research care and pioneering a unique and novel opportunity in transitional care.

This database will help us: 1. To develop and revise (as necessary) standards of care and treatment best practices for patients transitioning to adolescents with congenital genitourinary malformation. 2. To share evidence-based information between physicians across the country, advancing best practices for the secondary conditions of spina bifida, exstrophy, neurogenic bladder and bowel, and hydrocephalus. 3. To implement benchmarks to improve care in transitional urology clinics. 4. Evaluate the clinical cost-effectiveness of care offered.

ELIGIBILITY:
Inclusion Criteria:

- Primary diagnosis of congenital genitourinary abnormality leading to neurogenic bladder such as myelomeningocele, exstrophy, cerebral palsy, posterior urethral valve, congenital cardiac anomalies, chromosomal abnormalities, etc.

Exclusion Criteria:

- Non congenital neurogenic bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in Houston Methodist transitional urology clinic with congenital genitourinary abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-08-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life changes | 2 years
  The questionnaire is generated to collect long-term data regarding patients' genitourinary status including quality of life, kidney function, urine and fecal continence, sexuality, fertility, and pelvic health. Follow up information will be collected at baseline and 12 months follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No